CLINICAL TRIAL: NCT00549380
Title: A Clinical Study of Aneurysm Exclusion Using Endologix, Inc. Endoluminal Technology
Brief Title: Clinical Study of Aneurysm Exclusion
Acronym: Endologix
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arizona Heart Institute (Other)
Responsible Party: Edward B. Diethrich, MD, Arizona Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G990189
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Aneurysm
Keywords: Aneurysmal Disease in Thorax, Abdominal or Extremity
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Endologix, Inc. Endoluminal Technology

INTERVENTIONS:
Device: Endologix, Inc. Endoluminal Technology — Stent-graft endoprosthesis is inserted by Delivery System via a surgical cutdown (e.g., external iliac artery, femoral artery, common iliac artery conduit, etc.) approach. The insertion method depends on each patient's anatomy and is determined by the Clinical Investigator.

SUMMARY:
The ultimate purpose is to explore potential techniques to exclude aneurysms and provide alternative conduit for arterial flow. The single center sponsorship is intended to provide the investigators the potential to incorporate improvements in existing technology during the course of the study thereby ultimately enhancing the potential for superior medical care of patients suffering from these disease states.

DETAILED DESCRIPTION:
The primary objective of this study is to examine the feasibility of expanded applications of the basic Endologix technology for the treatment of arterial aneurysmal disease. A second objective of this study is to gather data in order to make logical, scientific recommendations for device design, construction and application which will expand the application of the endoluminal graft technology and improve its safety and efficacy while expanding the several potential future positive aspects of a less invasive method of treating arterial occlusive disease.

Endologix, Inc. has applied for and received an IDE for the investigation of a bifurcated device to exclude aneurysms of the abdominal aorta. The Arizona Heart Institute experience indicates that this small study design will prove successful. Using the basic technology of the current approved IDE, it is Arizona Heart Institute's intention to expand the scope of application and design in order to address a greater population basis suffering from aneurysmal disease. In this regard, the basic Endologix device designs will be applied to appropriate patients beyond the scope of the current bifurcated IDE. Patients meeting the criteria for the Endologix IDE will be enrolled independently in that study and followed precisely in order to comply with the study design. Patients with aneurysmal disease not currently filling the criteria for a bifurcated abdominal aortic prosthetic but who could potentially benefit from the technology to exclude aneurysmal disease will be considered from this study.

The patient's participation in the Study will include enrollment, Investigational Device procedure and follow-up period. Patient data will be collected for 1, 6, and 12 months and beyond as indicated. Subject follow-up at 1 month will include; ABIs, a complete Physical Examination, Duplex Ultrasound, and X-ray. Subject follow-up at 6 and 12 months will also include ABIs, a complete Physical Examination, CT Scan-Contrast Enhanced (unless contraindicated), CT Scan-No Contrast, and X-ray.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Informed consent understood and signed.
* Compliance with post-treatment follow-up requirements.
* Candidates in this study may not be ideal surgical patients and therefore may be included based upon the recommendation of the principal investigator or co-investigators and one independent consultant confirming the opinion of the investigators.
* Patient may present as an emergency or urgent use patient with indications including: ruptured aneurysm, dissected artery, or transected artery.

Exclusion Criteria:

* Life expectancy < 2 years.
* Pregnant or lactating women.
* Indication that appropriate follow-up studies would for whatever reason be difficult to obtain.
* Patient has other medical or psychiatric problems, which in the opinion of the investigator, precludes them from participating in the study.
* Anticoagulation drugs are indicated.
* Coagulopathy or bleeding disorder.
* Active systemic or localized groin infection.
* Inferior mesenteric artery is indispensable.
* Creatinine level > 1.7 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 1999-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility applications | Index procedure and discharge following index procedure
  The primary objective of this study is to examine the feasibility of expanded applications of the basic Endologix technology for the treatment of arterial aneurysmal disease.

SECONDARY OUTCOMES:
Data collection | 1 month
  A secondary objective of this study is to gather data in order to make logical, scientific recommendations for device design, construction, and application which will: a) expand the application of the endoluminal graft technology and b) improve its safety and efficacy while c) expanding the several potential future aspects of a less invasive method of treating arterial disease.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States